CLINICAL TRIAL: NCT02327884
Title: Characterization of Diseases With Salivary Gland Involvement
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150051; 15-D-0051
Record Dates: First submitted 2014-12-30; First posted 2014-12-31 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Healthy Volunteer; Sjogren's Syndrome; Salivary Gland Disease
Keywords: Genetics; Dry Mouth; Sjogren's Syndrome; Gland dysfunction; Induced Pluripotent Stem (iPS) Cell Lines
MeSH Terms: conditions — Sjogren's Syndrome; Salivary Gland Diseases; Xerostomia; Ichthyosis prematurity syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Healthy Volunteers matched with Sjogren's Syndrome patients
- Group 2: Family Members, affected and unaffected
- Group 3: any other cause salivary gland dysfunction

SUMMARY:
Background:

- Salivary glands in and around the mouth and throat make saliva. Salivary gland disorders can affect a person s quality of life. Studying people who have a disease that affects their salivary gland(s) may teach researchers about the disorders and their genetics.

Objectives:

- To study salivary gland diseases and disorders. To collect data and samples from people with salivary gland problems and their relatives.

Eligibility:

* People more than 4 years old who have or are suspected to have a disease involving salivary glands.
* Their relatives more than 4 years old.
* Healthy volunteers 18 years or older.

Design:

* Participants may be screened with:
* Medical history
* Physical exam
* Blood and urine tests
* General oral and dental history and exam
* Saliva collection
* Eye exam and test for dry eyes
* Health questionnaires (adults)
* Biopsy of some minor salivary glands. A small incision will be made on the inside of the lower lip and several tiny salivary glands will be removed.
* Participants will have 2-3 visits. These may include:
* Repeats of some screening tests
* Ultrasounds of some glands. Researchers will put some gel on the face, then press on it with a smooth wand.
* Adults may have other biopsies
* A small catheter inserted into the opening of the parotid gland duct on the inside of the cheek. A saline solution (in a syringe) will fill the duct.
* Swishing a saltwater solution in the mouth for 10 seconds and then spitting into a cup
* Scrapings collected from teeth, tongue, and cheeks

DETAILED DESCRIPTION:
This protocol is intended to allow disease-specific investigations in subjects with presentations of diseases with salivary gland involvement and will enable the collection of data, biological fluids and tissue samples from those subjects, their family members and normal controls, in order to assist our studies of understanding salivary gland disease pathophysiology. The exocrine salivary glands, by secreting saliva, play a critical role in the homeostasis of the oral cavity, which is the initial part of the gastrointestinal track. Several diseases including Parkinson s and systemic amyloidosis can be diagnosed through biopsies of easily accessible salivary glands. Moreover, several drugs and systemic diseases cause salivary gland hypofunction through unknown mechanisms.

We may evaluate participants with complaints of dry mouth to determine the cause and severity of their salivary gland dysfunction and their possible eligibility for other NIDCR protocols. Salivary secretions have antibacterial, lubricating, remineralizing, digestive, buffering and cleansing properties. Impaired function of these glands can cause an increase in tooth decay; a variety of oral hard and soft tissue changes, with painful, burning or ulcerated or oral mucosa; problems chewing, swallowing and speaking; and diminished taste and smell.

This protocol will provide us with the opportunity to learn from a variety of pathologies that involve directly or indirectly the salivary glands, expand our knowledge about these disorders and provide access to patients of interest for research, teaching, and clinical experience. Information obtained through this protocol may lead to potential innovative therapeutic studies. In addition to its role in investigating individuals who are of interest to the Sjogren s syndrome (SS) and Salivary Gland Dysfunction Unit of the MPTB of NIDCR, this protocol can provide a possible avenue for enrolling subjects from other NIH programs or other NIH protocols that exhibit signs or symptoms associated with the salivary glands dysfunction.

Design:

This is a single-site, observational, natural history, definition of phenotype, genotype/phenotype correlation; prospective linkage/gene identification study. This study has three groups:

Group 1: Well-defined SS subject patients with matched adult healthy volunteers

Group 2: SS/other pathology-adults/minors patient subjects and affected and unaffected family members

Group 3: Subjects of interest with any cause for salivary gland dysfunction (adults and minors)

Outcome Measures:

Primary Endpoint:

This is primarily a hypothesis generating, descriptive study. This protocol will allow disease-specific investigations to enable the collection of data, tissue, saliva, and blood and urine samples on subjects, their family members and healthy controls, to assist in the understanding of disease pathophysiology.

Secondary Endpoints:

Mechanistic genetic and inflammatory endpoints will be studied to gain insight into the molecular mechanism of Sjogren's syndrome and other diseases related to salivary gland pathologies to generate hypotheses for future research. The mechanistic outcome measures may include, but will not be limited to, functional studies of epithelial and immune cells, various histologic measures and biomarker studies and generation of iPSC for future therapies. Summary statistics employed may include means, geometric means, minimum and maximum values, standard deviations, 90% confidence limits, medians, and frequencies as appropriate for the measure. Genomic and genetic studies will allow the exploration of genetic alterations that might cause or influence the studied salivary gland pathologies.

Exploratory Endpoints:

As above

ELIGIBILITY:
* INCLUSION CRITERIA:
* Persons older than 4 years of age, affected with or suspected of being affected with a disease/disorder involving the salivary glands or who is a relative of a person who is affected with these diseases/disorders.

Or,

- Persons 18 years or older with active hepatitis with or without sicca symptoms and patients undergoing immunotherapy with an immune checkpoint inhibitor for oral cancer.

Specific to patients undergoing immunotherapy with an immune checkpoint inhibitor for threatment of oral cancer, these patients will be seen before and after check point inhibitor therapy which will coincide with 4 weeks (+/-2 weeks) before and again immediately before (+/- 2 weeks) definitive oral cancer treatment initiation (e.g., surgical resection, etc.).

Or,

- Healthy persons age 18 or older, who agree to have blood, urine, saliva or tissue samples collected and studied.

EXCLUSION CRITERIA:

* Anyone not able to give consent/assent or parental/guardian consent
* NIH employees who report directly to the principal investigator
* Significant concurrent medical condition or other circumstances that may affect the participant s ability to tolerate or complete the study, such as concurrent chemotherapy or bleeding disorders.

  * Specific only to the immune checkpoint inhibitor patients, oral cancer as a serious concurrent medical condition, will not serve as an exclusion criteria.
  * Moreover, these immune checkpoint inhibitor subjects, if unable to tolerate the study procedures, such as salivary gland biopsies, saliva collections, and/or oral exams, will be excluded as determined by the Principal Investigator.
* Additional exclusion criteria for Healthy Volunteers (HV):

  * Pregnancy
  * Sicca Symptoms
  * HIV, hepatitis B or C infection
  * Chronic medical illness, other than well-controlled hypertension or hyperlipidemia
  * Chronic use of medications, with the exception of oral contraception, hormone replacement therapy, aspirin, antihypertensives and antilipemics

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with known or suspected Sjogren's syndrome and their family members (affected and unaffected) are potentially eligible participants. Subjects with other causes of salivary gland dysfunction (including hepatitis C) may also be potentially eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2015-04-03 (Actual); Primary Completion 2032-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
hypothesis generating | hypothesis generating
  hypothesis generating

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Beach, P.A.-C, Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This is an observational study that began enrolling in 2015. De-identified data will be made public consistent with NIH policies.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The time frame is at the time of publication or within a year of study completion.
Access Criteria: The information will be shared publicly. No restrictions.

REFERENCES:
- [Derived] Joachims ML, Khatri B, Li C, Tessneer KL, Ice JA, Stolarczyk AM, Means N, Grundahl KM, Glenn SB, Kelly JA, Lewis DM, Radfar L, Stone DU, Guthridge JM, James JA, Scofield RH, Wiley GB, Wren JD, Gaffney PM, Montgomery CG, Sivils KL, Rasmussen A, Farris AD, Adrianto I, Lessard CJ. Dysregulated long non-coding RNA in Sjogren's disease impacts both interferon and adaptive immune responses. RMD Open. 2022 Nov;8(2):e002672. doi: 10.1136/rmdopen-2022-002672. PMID 36456101
- [Derived] Yin H, Pranzatelli TJF, French BN, Zhang N, Warner BM, Chiorini JA; NIDCD/NIDCR Genomics and Computational Biology Core. Sclerosing Sialadenitis Is Associated With Salivary Gland Hypofunction and a Unique Gene Expression Profile in Sjogren's Syndrome. Front Immunol. 2021 Jul 30;12:699722. doi: 10.3389/fimmu.2021.699722. eCollection 2021. PMID 34400910
- [Derived] Tanaka T, Warner BM, Odani T, Ji Y, Mo YQ, Nakamura H, Jang SI, Yin H, Michael DG, Hirata N, Suizu F, Ishigaki S, Oliveira FR, Motta ACF, Ribeiro-Silva A, Rocha EM, Atsumi T, Noguchi M, Chiorini JA. LAMP3 induces apoptosis and autoantigen release in Sjogren's syndrome patients. Sci Rep. 2020 Sep 16;10(1):15169. doi: 10.1038/s41598-020-71669-5. PMID 32939030
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-D-0051.html